CLINICAL TRIAL: NCT03229928
Title: Clinical Testing of a Real-Time Behavior Measurement Tool: Measuring Outcomes for CHAnge
Acronym: MOCHA
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); RTI International (Other)
Responsible Party: Sponsor
Other Study IDs: 16-2083; 4DR61604 (Other: National Center for Advancing Translational Science)
Record Dates: First submitted 2017-07-19; First posted 2017-07-26 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Neurodevelopmental Disorders
Keywords: Behavior; Outcome Measures; Intellectual/Developmental Disabilities
MeSH Terms: conditions — Neurodevelopmental Disorders; Behavior; Developmental Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (3):
- Stakeholder Advisory Panel: The investigators will recruit 2 parents of children with IDD, 2 special education teachers, and 2 behavior health professionals to assist with the development and initial testing of the upgraded MOCHA application features to test usability.
  Interventions: Device: MOCHA
- Primary Participants: The study primarily involves recruitment of clinically referred minor patients with IDD and their parents and teachers. Parents and teachers of 10 patients with IDD and co-morbid behavior problems will be asked to collect data via the MOCHA application on the frequency, antecedents,consequences, and other correlates of specific behavioral concerns.
  Interventions: Device: MOCHA
- Sensor Wearing Participants: These will be the same participants from aim 2. All participants will be offered the opportunity to wear the sensors and provide and chose which ones they would prefer to wear. Two participants will be asked to wear the sensor for 48 hours in order to pilot test the feasibility of syncing sensor and MOCHA application data collection.
  Interventions: Device: MOCHA

INTERVENTIONS:
Device: MOCHA — * MOCHA phone-based application
  * Event tracker button that marks the beginning and end of a behavioral event. Similar to a FOB that connects to MOCHA application via bluetooth
  * Wrist based sensor (applicable only to sensor wearing participants).

SUMMARY:
The efficacy of clinical trials addressing behavioral issues in individuals with intellectual/developmental disabilities (IDD) has traditionally been hampered by lack of objective and sensitive measures. While there are many behavioral observation measures available, most of them either rely on recall of the event or are designed for use by trained professional observers, requiring a third party or extensive training for use. The Measuring Outcomes for CHange (MOCHA) phone based application was developed to address the need for feasible real-time tracking of behavior. For the current study, 2 parents of children with IDD, 2 special education teachers, and 2 behavior health professionals will be recruited to serve on a stakeholder advisory panel. These individuals will provide initial feedback on the use of the application. Primary participants will be the parents and teachers of 10 children or adolescents (age 5-17 years) who are seeking treatment and support for the child's challenging behaviors (aggression, self-injurious behaviors, severe irritability) from clinicians in the Behavior Medicine Clinic at the Carolina Institute for Developmental Disabilities. Participants in the study will use MOCHA to record the child's behavior each time it occurs over 6 weeks in order to test the feasibility of using MOCHA over time and in response to treatment. The first 2 weeks of data collection will occur prior to the participant's scheduled visit to the BMC. Following the clinic visit, where clinically determined treatment suggestions will be provided, participants will continue to collect data for 4 weeks to determine if long term data collection is feasible and if change can be detected in response to the treatment through MOCHA (and compared to pen and paper questionnaires). Two children will be chosen from this participant pool to wear a sensor device to determine feasibility of syncing wearable sensors with the MOCHA app for use in future research studies. Following the 6 weeks of MOCHA use, all participants will receive a call or in person visit to conduct an exit interview about the participant's experiences using MOCHA. The overall goal of this study is to determine the feasibility of the use of the MOCHA application to track behaviors in populations of children with IDD. The MOCHA app does not act as an intervention and is not modifying the environment of the participants, but will be used as a tool by caregivers to track behaviors in real time.

DETAILED DESCRIPTION:
Behavior problems occur frequently and are a persistent source of treatment needs in individuals with intellectual and developmental disabilities (IDD). Problem behaviors such as aggression, self-injurious behaviors (SIB), destruction of property, and irritability can result in harm to self or others, interfere with social relationships, disrupt important family processes, and compromise positive individual and family adaptation. The impact of problem behaviors can have long term impacts for the individual, including reduced exposure to education, reduced quantity and quality of social interactions, and increased likelihood of more restrictive learning and living environments. Individuals with IDD who exhibit severe aggression are more likely to be placed in residential treatment facilities and to be placed on antipsychotic medications. Challenging behaviors have also repeatedly been shown to be strongly associated with poorer mental and physical health in caregivers. While there is a long history of both behavioral and pharmacologic interventions for aggression and SIB, the evidence base is considered slim compared to other fields in health care. A key challenge for clinicians and researchers in the IDD field is determining the efficacy of treatments to meet the complex needs of their patients. The ability to adequately assess the efficacy of any pharmacological or behavioral treatment has been limited by the lack of objective, real-time measurement tools. While there are many measures of behavior, including behavioral observation tools designed to assess the frequency, severity, and functions of specific behaviors, these measures are often limited. Most behavior measures rely either on recall (e.g., parent rating scales), or trained observers who, in addition to requiring specific training in behavior observation techniques also, as a factor of their presence, may change the behaviors and/or outcomes. The limitations inherent in these traditional measurement techniques have at best made it difficult to test the true efficacy of a clinical intervention, and, at worst, potentially resulted in the failure of clinical trials for medications which may have shown positive results with more sensitive and objective outcome measures.

MOCHA was developed in response to these challenges as an innovative yet simple method to capture behaviors in real time. MOCHA is available for both iOS and android platforms and can be sent remotely via a link to an individual's phone. MOCHA allows parents or teachers to record a behavior event simply by opening an app on their phone or tablet. A series of questions about the event allow for a brief yet comprehensive description of the event for use in understanding potential antecedents and functions of the behavior. Data is securely uploaded to a remote server at RTI whenever the participant is online. MOCHA was originally developed and piloted through internal funding to Dr. Wheeler at RTI International. The pilot study of four parents and three teachers of children with IDD was conducted primarily to establish feasibility and acceptability data and to engage stakeholders in a user-centered design approach to the development of the tool. Results from the pilot suggest that MOCHA is an acceptable and feasible tool to capture behaviors during or shortly after a behavior event. All parents and teachers in the pilot endorsed that MOCHA was easy to learn, clear and understandable, easy to answer questions, easy to use and a useful tool. Participants also reported the ability to record the behaviors and answer all follow up questions either when the behavior occurred or shortly after. In order to optimize the potential for MOCHA as an outcome measure there is a need to test its utility for measuring behaviors over time and in response to treatment.

The aims for this next phase of feasibility of MOCHA are as follows:

Aim 1. Expand the current MOCHA application to include additional clinically relevant features. Several features were suggested by participants in the development study to improve the usability of MOCHA. Specifically, the ability to personalize the target behaviors ahead of data collection; the use of a sync-able, wearable external event marker (EEM); and a feedback feature with graphed data to assist with monitoring behavior over time were requested features. Fortunately, MOCHA was developed using the Personal Health Informatics Toolkit (PHIT), a RTI developed, configurable, mHealth platform for developing apps and facilitating research. The PHIT platform has been used successfully for other apps with features such EEM and physiological sensors, similar to the features the investigators are proposing. Further, RTI has become an international leader in clinical informatics and provides shared resources and access to experts through its iSHARE (Integrating Signals and Human Response) program. Capitalizing on these resources, our first goal will be to develop and integrate these proposed features, using user-centered design procedures and engaging stakeholders in development.

Aim 2. Test the use of the MOCHA application to measure change in behaviors over time and in response to intervention. In order to assess the ability to use MOCHA the investigators will provide MOCHA to 10 families of individuals with IDD who are receiving intervention services through an established behavioral medicine clinic. The primary purpose of this aim is to examine the feasibility of the MOCHA app for use in recording frequency, intensity, and occurrence of behaviors and considering that information with parent perception/report.

Aim 3. Explore the ability to sync MOCHA with physiological data via wearable sensors. An ultimate vision of the MOCHA system includes the ability for the app to provide "ground truth" observable behavior that occurs in conjunction with physiological changes. Although full testing of a syncable system is outside the budgetary and time restrictions of this funding mechanism, the investigators propose to move this vision closer to reality by a) identifying wearable sensors that are acceptable and tolerable to the population and b) testing the feasibility of time syncing physiological markers with MOCHA identified behaviors.

ELIGIBILITY:
Inclusion Criteria:

Individual being monitored through MOCHA

* Ages 5-17 years
* Documented intellectual/developmental disability
* Presentation of aggression, self-injurious behavior, pica, or similar behavioral challenges
* Has at least 1 parent who speaks English
* Seeking consultation with professionals through the Behavior Medicine Clinic at the Carolina Institute for Developmental Disabilities

Parent and teacher of individual being monitored through MOCHA

* Unlimited age range
* English speaking

Exclusion Criteria Individual being monitored through MOCHA - Those who do not have a caregiver who speaks English will be excluded due to lack of professionals and materials in other languages

Parent and teacher of individual being monitored through MOCHA

- Those who do not speak English

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population includes individuals with IDD who have been referred to the Behavior Medicine Clinic at the Carolina Institute for Developmental Disabilities.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
MOCHA Exit Interview Score | End of Treatment [or Study Period], approximately 6 weeks
  The MOCHA exit interview is a study developed survey used to better understand client usability of MOCHA. Questions include items measured on a Likert scale measuring range of agree-ability (Strongly Disagree [0] to Strongly Agree [5]), frequency (Never [0] to Very Often [4]), or likelihood of use (Very Unlikely [0] to Very Likely [5]) to a question prompt. Additional open-ended questions are also included. The investigators will present the mean score obtained on these interview questions and compare the number of individuals who fell above and below that score. Qualitative responses will be coded for themes and presented.

SECONDARY OUTCOMES:
MOCHA Use Frequency | End of Treatment [or Study Period], approximately 6 weeks
  Data from the MOCHA application will be extracted to determine the frequency of use. Mean scores will be presented.
MOCHA Clinician Interview Score | At Study Completion, approximately 5 months
  The MOCHA clinician interview is a study developed survey used to better understand clinician usability of MOCHA. Questions include items measured on a Likert scale measuring range of agree-ability (Strongly Disagree [0] to Strongly Agree [5]), frequency (Never [0] to Very Often [4]), or likelihood of use (Very Unlikely [0] to Very Likely [5]) to a question prompt. Additional open-ended questions are also included. The investigators will present the mean score obtained on these interview questions. Qualitative responses will be coded for themes and presented.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Mankowski, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Carolina Institute for Developmental Disabilities, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No